CLINICAL TRIAL: NCT00543816
Title: MK0767 Added to Insulin Therapy in Patients With Type 2 Diabetes (0767-030)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-030; 2007_628; MK-0767-030
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
This study will look to see if MK0767 works better than placebo in controlling blood sugar in patients with Type 2 Diabetes who are taking insulin but do not have adequate control of their blood sugar.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes with inadequate glycemic control
* Patient is on stable insulin therapy alone or with one oral antidiabetic agent
* Male or non-pregnant female 21 years or older
* Total daily dose of insulin must be less than or equal to 30 but not greater than or equal to 200 units/day

Exclusion Criteria:

* Have a history of type 1 diabetes mellitus
* History of ketoacidosis who are being treated with insulin
* Are taking 2 or more antidiabetic agents in combination with insulin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-08; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC